CLINICAL TRIAL: NCT04436913
Title: Evaluation of Prevention Potential of Preventive Regimens Containing Herbal-based and Fluoride-based Toothpastes Versus Fluoride Varnish and Fluoride Toothpaste Only in High Caries Risk Patients: A Randomized Clinical Trial
Brief Title: Evaluation of Preventive Regimens With Different Toothpastes vs Fluoride Varnish & Toothpaste in High Caries Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hoda Abdelmeguid Mohamed Fathy Ismail Sabry, Principal Investigator , Master degree student, Conservative Dentistry Department, Faculty of Dentistry, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Himalaya complete care
Record Dates: First submitted 2020-06-15; First posted 2020-06-18 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- preventive regimen using Herbal toothpaste(Himalaya) (Experimental): The regimen includes herbal toothpaste containing "Neem , Miswak , Babool and Pomegranate" (Himalaya Complete Care).
  Interventions: Other: Himalaya complete care toothpaste
- preventive regimen using Fluoride based toothpaste (Signal). (Experimental): Participants will be using fluoride-based toothpaste (Signal), (1450 ppm sodium fluoride)
  Interventions: Other: Signal toothpaste
- Fluoride toothpaste and fluoride varnish (Active Comparator): Participants will be using fluoride-based toothpaste (Signal), (1450 ppm sodium fluoride) and fluoride varnish
  Interventions: Other: Signal toothpaste and fluoride varnish

INTERVENTIONS:
Other: Himalaya complete care toothpaste — Herbal toothpaste as a part of a caries preventive regimen
  Arms: preventive regimen using Herbal toothpaste(Himalaya)
Other: Signal toothpaste — fluoride based toothpaste as a part of a caries preventive regimen
  Arms: preventive regimen using Fluoride based toothpaste (Signal).
Other: Signal toothpaste and fluoride varnish — application of fluoride varnish and using fluoride based toothpaste
  Arms: Fluoride toothpaste and fluoride varnish

SUMMARY:
This study will be conducted in order to determine the prevention effect of caries preventive regimen using herbal toothpaste and regimen using fluoride toothpaste versus fluoride toothpaste and fluoride varnish on the caries risk of patients with high caries risk.

DETAILED DESCRIPTION:
Dental caries is highly predominant worldwide. So, in addition to treating this caries, patients should be managed to avoid new caries. Preventive measures could be applied to the patients who are most expected to develop dental caries who are identified by caries risk assessment. Thus, effective caries risk assessment is essential to control new caries development.

Dental caries can be prevented by conducting appropriate measures; therefore, it is crucial to identify those who are most likely to have dental caries by caries risk assessment and giving them the essential preventive measures. Though some caries preventive measures have showed success in descriptive clinical trials, there is little information on their practicality with high caries risk groups in everyday usage.

Oral health is an essential part of general well being, people have used herbs in order to prevent dental diseases for centuries. In 2008 the Federal Council of Dentistry approved the use of medicinal plants for oral healthcare.

Medicinal plants can heal bacterial diseases as it is full of antimicrobial agents. They are becoming more popular than chemicals due to the side effects of synthetic antibiotics and the antibiotic resistance in microorganisms.

Studies propose that herbal extracts are highly effective against significant microorganism which cause dental caries like Streptococcus mutans. Herbal toothpaste decreases dental caries through combined effects of antibacterial agents, oral acid neutralisers and decreased plaque bacterial enzyme inhibitors present in the herbal toothpaste.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients with free medical history.
* Age range 15-50 years.
* Patients with high caries risk assessment due to increased cariogenic bacteria according to Cariogram.
* low fermentable carbohydrates diet patient
* Not under antibiotic therapy either at the time of the study or up to the last month before the start of the study.

Exclusion Criteria:

* Patients with a compromised medical history.
* Cariogenic diet patient.
* Extreme plaque accumulation and periodontal problems
* Participants with a history of allergy to any of the drugs or chemicals used in the study.
* Patients on any antibiotics during the past month

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2021-01-16 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Caries risk assessment | Outcomes will be evaluated at baseline, after 1 week, after 4 weeks and after 12 weeks.
  Change in caries risk assessment by "cariogram software" as each patient data is collected in order to be inserted into the "Cariogram software" which in turn will evaluate this data and lead to a pie chart showing the chance of avoiding new caries as percentage.
  This data includes caries experience, related diseases, diet content, fluoride program, salivary buffer capacity, saliva secretion rate, diet frequency, "Mutans streptococci" count, amount of plaque, and clinical examination.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Faculty of oral and dental medicine, Cairo, Egypt